CLINICAL TRIAL: NCT01871142
Title: Double-Blind, Placebo Controlled Evaluation of the Attenuation by Aes-103 of Hypoxia Mediated Decrements in Endurance Exercise Performance in Healthy Adult Humans
Brief Title: Evaluation of the Attenuation by Aes-103 of Hypoxia Mediated Decrements in Endurance Exercise Performance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: AesRx, LLC (Industry)
Responsible Party: Principal Investigator, Christopher Bell, Associate Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 13-4002H
Record Dates: First submitted 2013-05-29; First posted 2013-06-06 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Hypoxia
Keywords: 5 Hydroxymethyl 2 Furfural; AES103; Exercise
MeSH Terms: conditions — Hypoxia; Motor Activity | interventions — 5-hydroxymethylfurfural

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Randomized crossover assignment (Experimental): Participants will receive, in a random order, a placebo prior to exercise in normoxia, a placebo prior to exercise in hypoxia, 1000 mg of Aes-103 prior to exercise in hypoxia, and 3000 mg of Aes-103 prior to exercise in hypoxia. Each intervention is separated by a 7 day washout period.
  Interventions: Drug: Placebo; Drug: Aes-103

INTERVENTIONS:
Drug: Placebo — 100 mL
  Other Names: Tropicana Pure Premium Orange Juice
Drug: Aes-103 — Single dose of 1000mg Aes-103 dissolved in 100 mL of Tropicana Pure Premium Orange Juice
  Other Names: 5-Hydroxymethyl-2-Furfural (5-HMF)
Drug: Aes-103 — Single dose of 3000mg Aes-103 dissolved in 100 mL of Tropicana Pure Premium Orange Juice
  Other Names: 5-Hydroxymethyl-2-Furfural (5-HMF)

SUMMARY:
In low oxygen environments, such as high-altitude, some adults may become ill and suffer from acute mountain sickness. Further, all adults will find that exercising becomes much more difficult when compared with exercise at lower altitudes (e.g. sea-level). The purpose of this investigation is to study the effects of a new medicine called Aes-103. A company called AesRx, LLC makes this medicine. The active ingredient in the medicine is 5-Hydroxymethyl-2-Furfural (5HMF), a naturally occurring substance that can be found in coffee, honey, dried fruits, fruit juices, malt, barley, Balsamic vinegar and caramel.The investigators believe that Aes-103 may help people adjust to high-altitude quickly and prevent them from becoming ill. The purpose of the study is to determine if Aes-103 will promote endurance performance in low oxygen environments in healthy adult humans.

Aes-103 is currently being investigated by AesRx, LLC (Newton, MA) in collaboration with the National Heart, Lung and Blood Institute of the NIH (Bethesda, MD) as a potential anti-sickling agent in sickle cell disease. Sickle-cell disease is characterized by problems in blood that prevent blood cells from carrying oxygen. Aes-103 might be able to help blood cells carry more oxygen. It is for this reason that the investigators in this study believe Aes-103 might help people adjust to high-altitude quickly.

There are no known special safety considerations with the active ingredient in Aes-103 (5-HMF). In recent, placebo controlled, clinical safety tests, Aes-103 was given in single doses of 300 mg, 1000 mg,2000 mg and 4000 mg to healthy normal volunteers. Additionally, the toxicological effects of Aes-103 have been studied when given acutely, sub-acutely, and chronically in rodents, and for up to 28 days in dogs. Based on these safety studies, single doses of Aes-103 are expected to have no significant negative/toxicological effect at the doses being evaluated in this study.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind blind, repeated measures (cross-over) study. Approximately 12 healthy adult men will consume, in a random order, a placebo prior to exercise in normoxia, a placebo prior to exercise in hypoxia, 1000 mg of Aes-103 prior to exercise in hypoxia, and 3000 mg of Aes-103 prior to exercise in hypoxia.

Study participants will report to the Human Performance/Clinical Research Laboratory (HPCRL) on 6 separate occasions. On visit 1 study participants will undergo screening (e.g. medical history and 12-lead electrocardiogram and blood pressure at rest and during incremental exercise to volitional exhaustion), and will be instructed to avoid foods and drinks high in 5-HMF (e.g., coffee, malt, barley, dried fruits, and caramel) for at least 3 days before each subsequent visit. Visit 2 will comprise of a habituation visit during which subjects will be given the opportunity to rehearse the exercise test. Visits 3, 4, 5 and 6, will occur in a random order and be almost identical in nature. Study participants will abstain from vigorous physical exercise and alcohol consumption during the 24-hours prior to each visit. In addition, study participants will abstain from all food and beverages, except water, during the 4-hours prior to visits 3, 4, 5 and 6. On arrival subjects will be instrumented for measurement of heart rate, blood pressure and blood oxygen saturation. Following baseline determination subjects will consume either: a placebo, 1000 mg of Aes-103 or 3000 mg of Aes-103. 45 minutes after consumption, participants will enter our environmental chamber, adjusted randomly to either normoxia (21% oxygen) or hypoxia (15% oxygen). The pairing of normoxia/hypoxia and supplement will be as follows: placebo + normoxia, placebo + hypoxia, 1000 mg + hypoxia, and 3000 mg + hypoxia. Participants will remain seated in the environmental chamber for 15 minutes, after which they will complete a standardized warm-up bout of exercise (100 W for 30 minutes) followed by a brief time trial (time taken to cycle 12.5 km (~7.75 miles)). Heart rate, blood pressure and blood oxygen saturation will be recorded every 5 minutes. During exercise, subjective ratings of perceived exertion (Borg Scale) will be recorded every 10 minutes, and at end-exercise.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male volunteer, aged 18-40 years old, body mass index 18-30 kg/m2, inclusive
* Have successfully completed a screening visit consisting of medical history, physical examination, 12-lead ECG, blood pressure, blood oxygen saturation at rest and during incremental exercise to volitional exhaustion (Note: Subjects with abnormal screening values may be eligible if the results are not clinically significant, as judged by the investigator or medical monitor)
* Be able to understand and have provided written informed consent including signature on an informed consent form approved by an institutional review board
* Have provided written authorization for use and disclosure of protected health information
* Agree to abide by the study schedule and dietary restrictions and to return for the required assessments
* Be willing to abstain from foods high in 5-HMF (e.g., coffee, malt, barley, balsamic vinegar, dried fruits,and caramel products) for at least 3 days prior to each dosing
* Be willing and able to repeatedly perform exhaustive cycle ergometer exercise

Exclusion Criteria:

* Have evidence of clinically significant cardiovascular, respiratory, renal, hepatic, pulmonary, gastrointestinal, hematological, neurological, psychiatric, or other disease that may interfere with the objectives of the study or the safety of the subject, as judged by the investigator in agreement with the sponsor or medical monitor, have been hospitalized in the past 2 years as a result of these conditions, or are receiving pharmacological treatment for these conditions
* Have taken prescription drugs or herbal preparations in the 2 weeks before dosing
* Is currently enrolled in another clinical study for another investigational drug or has taken any other investigational drug within 30 days before the screening visit
* Habitual and/or recent use of recreational drugs, such as cocaine, marijuana, opiates, amphetamines, methamphetamines, benzodiazepines,
* Have taken disulfiram, 4-methylpyrazole, or any other drug that is an inhibitor of alcohol dehydrogenase or aldehyde dehydrogenase within the past 30 days
* Have engaged in strenuous physical activity within 24 hours prior to dosing
* Be considered not suitable for participation in this trial for any reason, as judged by the investigator

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bell, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

REFERENCES:
- See also: Department of Health and Exercise Science, Colorado State University — http://www.chhs.colostate.edu
- See also: Initial Safety Trial For Treatments Under Investigation In Current Study — http://www.clinicaltrials.gov/ct2/show/NCT01597401?term=Aes-103&rank=1

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Randomized Crossover Assignment
Started | 12
Received Placebo + Normoixa | 11
Received Placebo + Hypoxia | 12
Received 1000mg Aes 103+ Hypoxia | 11
Received 3000mg Aes-103 + Hypoxia | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed for all subjects that completed study.
Groups:
- Entire Study Population: All enrolled participant baseline data
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 12
Height [Mean (Standard Deviation); unit: meters] | 1.75 (0.03)
Body Mass (kg) [Mean (Standard Deviation); unit: Kilograms] | 74.8 (6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (2)
Fat Mass (kg) [Mean (Standard Deviation); unit: kilograms] | 14.1 (4)
Lean Mass (kg) [Mean (Standard Deviation); unit: kilograms] | 56.7 (5)
Percent Body Fat [Mean (Standard Deviation); unit: Percentage of body fat] | 19 (4)
Waist Circumference (cm) [Mean (Standard Deviation); unit: centimeters] | 79.3 (5)
Waist-to-Hip Ratio [Mean (Standard Deviation); unit: ratio] | 79.3 (0.04)
Maximal oxygen uptake (VO2max (L/min)) [Mean (Standard Deviation); unit: Liters/minute] | 3.96 (0.06)
VO2max (ml/kg/min) [Mean (Standard Deviation); unit: milliliter/kilogram/minute] | 53.2 (8)
Maximal heart rate (HRmax (beats/min)) [Mean (Standard Deviation); unit: Beats/minute] | 187 (4)
Maximal respiratory exchange ratio (RERmax) [Mean (Standard Deviation); unit: VCO2/VO2] | 1.09 (0.02)

OUTCOME MEASURES:

1. Primary Outcome: Primary Objective Endurance Exercise Performance
Description: To quantify endurance exercise performance (time trial performance during stationary cycle ergometer exercise) in healthy adult men in four conditions: normoxia (normal oxygen; fraction of inspired oxygen = 0.21) following oral placebo consumption, hypoxia (low oxygen; fraction of inspired oxygen = 0.15) following oral placebo consumption, hypoxia following oral consumption Aes-103 (1000 mg) and hypoxia following oral consumption Aes-103 (3000 mg).
Time Frame: The time trial will begin after 1 hour after consumption of the intervention or placebo under normoxic or hypoxic conditions.
Measure: Mean (Standard Error); unit: minutes
Groups:
- Palcebo + Normoxia: Randomized crossover assignment for each participant. Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Normoxia (21% oxygen)
- Placebo + Hypoxia; 1000mg Aes-103 + Hypoxia; 3000mg Aes-103 + Hypoxia: Randomized crossover assignment for each participant.
  Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Hypoxia (15% Oxygen)
Arm/Group | Palcebo + Normoxia | Placebo + Hypoxia | 1000mg Aes-103 + Hypoxia | 3000mg Aes-103 + Hypoxia
Number analyzed (Participants) | 11 | 11 | 11 | 11
minutes | 22.4 (0.7) | 24.5 (0.5) | 24.0 (0.7) | 24.6 (0.6)

2. Secondary Outcome: Secondary Objective Safety and Tolerability
Description: To assess the safety and tolerability of single, escalating oral doses of Aes-103 compared with placebo in healthy adult men at rest and during stationary cycle ergometer exercise in normoxia and hypoxia by monitoring adverse events (AEs), electrocardiograms (ECGs), blood pressure, blood oxygen saturation.
Time Frame: AEs will be monitored at the time of visit and during the follow up period of 7 to 14 days.
Measure: Number; unit: participants
Groups:
- Placebo + Normoxia: Number of participants receiving placebo in normoxic conditions. Randomized crossover assignment for each participant. Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Normoxia (21% oxygen)
- Placebo + Hypoxia: Number of participants receiving placebo in hypoxic conditions Randomized crossover assignment for each participant. Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Normoxia (21% oxygen)
- 1000mg Aes-103 + Hypoxia: Number of participants receiving 1000mg Aes-103 in hypoxic conditions Randomized crossover assignment for each participant. Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Hypoxia (15% oxygen)
- 3000mg Aes-103 + Hypoxia: Number of participants receiving 3000mg Aes-103 in hypoxic conditions Randomized crossover assignment for each participant. Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Hypoxia (15% oxygen)
Arm/Group | Placebo + Normoxia | Placebo + Hypoxia | 1000mg Aes-103 + Hypoxia | 3000mg Aes-103 + Hypoxia
Number analyzed (Participants) | 11 | 12 | 11 | 12
participants | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Placebo + Normoxia: Participants receiving placebo in normoxic conditions Randomized crossover assignment for each participant. Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Normoxia (21% oxygen)
- Placebo + Hypoxia: Participants receiving placebo in Hypoxic conditions Randomized crossover assignment for each participant Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Hypoxia (15% Oxygen)
- 1000 mg Aes-103 + Hypoxia: Participants receiving 1000mg Aes-103 in hypoxic conditions Randomized crossover assignment for each participant. Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Hypoxia (15% oxygen)
- Hypoxia 3000 mg Aes-103 + Hypoxia: Participants receiving 3000mg Aes-103 in hypoxic conditions Randomized crossover assignment for each participant. Intervention 1 dose. Next random crossover assignment was followed by a 7 day washout period.
  Note: Hypoxia (15% oxygen
Arm/Group | Placebo + Normoxia | Placebo + Hypoxia | 1000 mg Aes-103 + Hypoxia | Hypoxia 3000 mg Aes-103 + Hypoxia
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/11 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Normoxia (N=11) | Placebo + Hypoxia (N=12) | 1000 mg Aes-103 + Hypoxia (N=11) | Hypoxia 3000 mg Aes-103 + Hypoxia (N=12)
Nausea leading to vomiting (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — During the participants first exposure to hypoxia, following consumption of 3 g of Aes-103, the participant reported feeling nauseous and light-headed prior then vomited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No